CLINICAL TRIAL: NCT02034396
Title: Clinical Implications of Genetic Variations of Venous Stasis Ulceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rabih A. Chaer, MD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PRO10120155
Record Dates: First submitted 2014-01-02; First posted 2014-01-13 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Venous Ulcers
Keywords: Ulcers, venous, unna's boot
MeSH Terms: conditions — Varicose Ulcer; Ulcer | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood draw (Other): One blood draw at enrollment
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — One blood draw at enrollment

SUMMARY:
Currently, there is no standard approach for the treatment of patients with venous stasis ulcers, and no means of accounting for the genetic factors that may contribute to a patient's response to different therapeutic interventions. In order to determine whether, or to what extent, genetic profiling of venous stasis ulcers can stratify patients according to their potential for disease progression or healing, and guide preventive strategies and levels of therapeutic interventions, the study will involve retrospective genetic profiling of patients with a healed or persistent venous stasis ulcer as a means of determining the efficacy of current therapies, and to establish a future prospective evaluation of treatment algorithms based on genetic phenotype and variation. Results obtained from the 2 aforementioned groups of participants will be compared with those of a control group of participants who have no history of venous ulcer nor peripheral vascular disease.

.

DETAILED DESCRIPTION:
A blood specimen will be drawn, medical and medication history taken, and wound/s will be assessed and followed for 2 years in regard to the enrollees w/active venous ulcer/s or healed venous ulcer/s.

A venous duplex ultrasound of right and left lower extremities will be done at no cost, a blood specimen will be drawn, and medical and medication history will be taken in regard to control group enrollees.

ELIGIBILITY:
Group 1-Active venous ulcer (CEAP 6) & Group 2-Healed venous ulcer (CEAP 5)

Inclusion Criteria:

* >/=18y.o.
* active venous ulcer (CEAP 6)
* healed venous ulcer (CEAP 5)

Exclusion Criteria:

* <18 y.o.
* inability to comply w/compression therapy
* Inability to maintain f/u schedule
* ABI (ankle-brachial index) < 0.5 if pedal pulses are not palpable
* Inability to ambulate w/active ulcer (N/A for Group 2)
* Diabetic w/ABI <0.5
* Severe premorbid systemic disease such as pulmonary failure, heart failure, renal failure, or hepatic failure w/a life expectancy of <1 year
* Chronic steroid therapy Group 3-Controls

Inclusion Criteria:

* >/= 50y.o.
* no reported clinical symptoms of venous disease
* (CEAP 0 or 1)

Exclusion Criteria:

* <50y.o.
* ABI (ankle-brachial index) < 0.5 if pedal pulses are not palpable
* Diabetic w/ABI < 0.5
* Severe premorbid systemic disease such as pulmonary failure, heart failure, renal failure, or hepatic failure w/a life expectancy of <1 year
* Chronic steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Ulcer healing | Assessment made when batch of samples (360) obtained
  Time to ulcer healing
Ulcer recurrence | Assessment made when batch of samples (360) obtained
  Presence of ulcer recurrence

SECONDARY OUTCOMES:
Analysis of genetic variation in concert with ulcer healing, time to healing and recurrence | Assessment made when batch of samples (360) obtained

OTHER OUTCOMES:
Analysis of association between clinical variables and genetic testing results | Assessment made when batch of samples (360) obtained
Analysis of clinical variables in conjunction with ulcer healing and recurrence | Assessment made when batch of samples (360) obtained

CONTACTS AND LOCATIONS:
Overall Officials: Rabih Chaer, MD, Principal Investigator — UPMC/UPP Vascular Surgery
Locations (1):
- UPMC Heart and Vascular Institute - Division of Vascular Surgery, Pittsburgh, Pennsylvania, United States